CLINICAL TRIAL: NCT02932657
Title: Perceived Impact of Art Therapy in Patients With Cystic Fibrosis (Adolescents, Adults and Transplanted Not Transplanted) and in Professional Interdisciplinary Teams Taking Care of Them.
Brief Title: Perceived Impact of Art Therapy in Patients With Cystic Fibrosis and in Professional Interdisciplinary Teams Taking Care of Them.
Acronym: MUCO-ART-PLUS
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC16_0285
Record Dates: First submitted 2016-10-12; First posted 2016-10-13 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Non interventional study — First individual interviews will be set up with teenagers of Nantes University Hospital . Then, focus group will be conduct with patients and professionals in Nantes and Foch University Hospital.

SUMMARY:
Cystic fibrosis is so far a disease whose treatment remains essentially symptomatic care teams perceive the boundaries of a support mainly focused on drug treatments. The patient had no other choice but to learn to live with their disease, the goal is to make every effort so that tames the disease while maintaining high self-esteem that gives meaning to his life, allowing, among other things, a good grip of treatment.

Through this research we hope to encourage the integration of art therapy in the course of care of cystic fibrosis patients, from children to adults before and after transplantation, in connection with the patient education and counseling

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis aged adolescents 13 to 18 years, as part of their monitoring at cystic fibrosis center of Nantes
* Adults over 18 years nontransplanted in their follow at cystic fibrosis center/transplantation center of Foch
* More than 18 adult transplant as part of their monitoring at cystic fibrosis center/transplantation center Foch
* Professional interdisciplinary teams taking care of the cystic fibrosis children center of Nantes, cystic fibrosis center/transplantation center of Foch
* Agreeing to participate in research

Non Inclusion Criteria:

* Patient refusal of adolescent parents to participate in the study
* Professional refusal of teams to participate in the study

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Will be included in this research project:
  * Adolescents aged 13 to 18, followed by the cystic fibrosis Children center of Nantes that have benefited from art therapy session
  * Non transplanted adult patients followed cystic fibrosis center of Foch and having already benefited from art therapy session
  * The transplanted adult patients followed the transplantation center Foch and having already benefited from art therapy session
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2018-01-28 (Actual); Study Completion 2018-01-28 (Actual)

PRIMARY OUTCOMES:
Patient responses to the effects of art therapy and music therapy | 1 day
  The depth interviews with patients will achieve a thematic and structural analysis of the speech. This will capture the effects of art therapy and music therapy on patients, their point of view.

CONTACTS AND LOCATIONS:
Overall Officials: Valérie David, Dr, Principal Investigator — Nantes University Hospital
Locations (2):
- France (2):
  - Nantes University Hospital, Nantes
  - Foch Hospital, Suresnes

IPD SHARING:
Plan to Share IPD: No